CLINICAL TRIAL: NCT02549742
Title: Electrochemotherapy on Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Irene Wessel, Consultant, ph.d., associate professor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH1222
Record Dates: First submitted 2015-09-06; First posted 2015-09-15 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Head Neck Cancer
Keywords: Electrochemotherapy; head neck cancer; bleomycin
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Electrochemotherapy; Electroporation; Drug Therapy; Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Electrochemotherapy (Experimental): 25 patients treated with electrochemotherapy
  Interventions: Procedure: Electrochemotherapy; Device: Cliniporator; Drug: Bleomycin

INTERVENTIONS:
Procedure: Electrochemotherapy — Electroporation by a device, Cliniporator, combined with chemotherapy, Bleomycin.
  Other Names: electroporation with chemotherapy; eletropermeabilization with chemotherapy
Device: Cliniporator — Electric pulses , duration 100 microseconds, about 400 V given at 5000 Hz.
Drug: Bleomycin — Administered intravenously or injected into the tumour before electroporation.

SUMMARY:
A phase II clinical trial testing electrochemotherapy on mucosal recurrent head and neck cancer. Twenty-five patients will be treated. Primary outcome is tumour response on imaging. Secondary outcomes are response from tissue samples, VAS score, Quality of life evaluation and side effects to treatment.

DETAILED DESCRIPTION:
Electric pulses may be used to transiently permeabilise cell membranes, enabling passage of otherwise non-permeating molecules. This dramatically enhances the cytotoxic effect of certain chemotherapeutic agents, and is termed electrochemotherapy. Electrochemotherapy is now standardly used in the treatment of cutaneous metastases of various cancers in over 100 cancer centers around Europe.

The intention of this trial is to investigate the possible use of electrochemotherapy in recurrent head and neck cancer as a palliative treatment. Surgery and radiotherapy, with the possible addition of chemotherapy, cures a large part of patients with head and neck cancer. However, in the event of recurrence curative options may be exhausted and the patient is referred for palliative chemotherapy.

It is for this patient group, the investigators propose electrochemotherapy in a clinical trial.

The electrochemotherapy is administered as a once-only treatment, with possible retreatment after eight weeks. Under general anesthesia, chemotherapy is administered intravenously, followed by application of electric pulses to the tumour area. Before treatment, the location and spread of the tumour is determined by imaging.

The trial includes evaluation of response by MRI (magnetic resonance imaging) and PET/CT (Positron Emission Tomography - Computed Tomography) scans (base-line, 4 weeks, 8 weeks), tissue samples, as well as adverse events registration and questionnaires on quality of life. The planned study is a phase II clinical study, prospective, observational with up to 25 patients.

Treatments will be performed in collaboration between the Department of Oncology, Copenhagen University Hospital Herlev, which has extensive experience in electrochemotherapy, and the Department of Ear Nose and Throat Surgery at Copenhagen University Hospital Rigshospitalet, that has the surgical expertise and set-up needed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age > 18 years.
2. Verified cancer of the head and neck area of any histology.
3. At least one tumour lesion should be accessible for electroporation.
4. Performance status WHO <= 2nd
5. Progressive and / or metastatic disease.
6. Expected survival of > 3 months.
7. Measurable disease is defined as at least one measurable lesion by RECIST 1.1.
8. A treatment-free interval of more than 4 weeks since chemotherapy or radiation therapy.
9. The participant should have been offered the current standard treatment. If there are no further standard treatment to offer or if the participant does not want to receive this, the participant may be included in the trial.
10. The participant should be able to understand the information for participants and be willing and able to comply with hospitalization in the treatment and the agreed follow-up visits and tests.
11. Platelets ≥ 50 billion / L, INR (international normalized ratio) > 1.5. Medical correction is permitted, e.g. correction using vitamin K.
12. Sexually active women who can become pregnant should use adequate contraception during this trial and 6 months after administration of bleomycin (pill, spiral, injection of prolonged progestin subdermal implantation, hormone-containing vaginal devices, transdermal patches).
13. Signed informed consent. -

Exclusion Criteria:

Participants should be excluded if they meet just one of the criteria stated below.

1. Symptomatic progression of the participants cancerous disease that requires another intervention.
2. Acute lung infection
3. Symptoms of lung function impairment. This triggers a lung function test (DLCO = diffusing capacity of the lungs for carbon monoxide), if moderate to severe the participant will be excluded.
4. Previous bleomycin treatment with cumulative dose more than 240,000 Units / m2.
5. History of severe allergic reactions associated with bleomycin.
6. Allergy to constituents of the planned anesthetic.
7. Coagulation disorder which can not be corrected.
8. Chronic renal dysfunction with creatinine> 150 micromoles / liter, will trigger a Cr-51-EDTA (Chromium-51-ethylenediamine tetra acetic acid) clearance. If this is too impaired, the participant is excluded.
9. Pregnancy or lactation.
10. While participation in other clinical trials involving experimental drugs or involved in a trial within 4 weeks prior to study drug administration.
11. Other disorders investigator finds incompatible with participation in the trial. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-02; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Tumour response from PET/CT scans (Positron Emission Tomography - Computed Tomography) | 8 weeks after treatment

SECONDARY OUTCOMES:
Tumour response from MRI scans (Magnetic resonance imaging) | 8 weeks after treatment
Tumour response from tissue samples | 4 weeks after treatment
  Still cancer activity or not
VAS score (Visual Analogue Scale) | baseline, 4 weeks and 8 weeks after treatment
  Participant assessed
Quality of life | baseline, 4 weeks and 8 weeks after treatment
  EORTC scores for head and neck (The European Organisation for Research and Treatment of Cancer)
CTCAE recordings (Common Terminology Criteria for Adverse Events) | baseline, 4 weeks and 8 weeks after treatment
  side effects scored by CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, MD, Study Chair — Denmark: Herlev and Gentofte Hospital, University of Copenhagen
Locations (1):
- Department of Otorhinolaryngology, Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided